CLINICAL TRIAL: NCT03441074
Title: Effects of Odor Enrichment on Delayed Neurocognitive Recovery
Brief Title: Olfactory Function and Delayed Neurocognitive Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Chief of Psychiatry, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: dsyy003
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Delayed Neurocognitive Recovery

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomly assigned to intervention group will get odor enrichment during the perioperative period
  Interventions: Behavioral: Odor Enrichment
- Non-intervention Group (No Intervention): Patients randomly assigned to non-intervention group will not get any odor enrichment during the perioperative period

INTERVENTIONS:
Behavioral: Odor Enrichment — Patients in intervention group will get odor enrichment during perioperative period (3 days before the surgery and 7 days after the surgery). Odor-enriched participants were exposed daily for 24 hours to different aromatic fragrances (phenyl ethyl alcohol - rose; eucalyptol - eucalyptus; citronellal - lemon; eugenol - cloves) referred to previous studies. Odors were changed for each subject after 24 hours. According to previous studies, 10 drops of the 100% essential oil (0.5 ml) were dropped on a fabric which was placed in tea bags hanging at the hospital bedside.
  Arms: Intervention Group

SUMMARY:
To explore whether odor enrichment can reduce the risk of delayed neurocognitive recovery as an intervention strategy.

DETAILED DESCRIPTION:
Postoperative neurocognitive disorder, one of the most common postoperative complications in older adults, includes acute postoperative delirium, delayed neurocognitive recovery (within the 30 days recovery period, dNCR), and postoperative neurocognitive dysfunction (from expected recovery 30 days to 12 months). Previous studies showed that the incidence of dNCR ranged from 18% to 40% and is mainly characterized by cognitive impairment, which can develop into long-term cognitive impairment, even elevating the risk of Alzheimer's Disease (AD) related dementia and premature mortality. These symptoms can have significant adverse effects on quality of life and may increase the risk of other physical and psychological disorders, potentially impacting social stability. These statistics underscore the importance of early detection and timely intervention in mitigating the long-term effects of dNCR. Despite the significance of dNCR, effective treatment options remain elusive.

Based on these insights, previous studies have explored the impact of olfactory enrichment in animal models. Zhang et al. demonstrated that surgery and anesthesia could cause olfactory impairment, which might contribute to dNCR, while suggesting that odor enrichment, a non-pharmacological intervention, could reduce postoperative cognitive impairment in animal models. Olfactory enrichment, also known as olfactory training, is a safe and affordable treatment and may have preventative or supportive effects on olfactory function or cognitive function. Evidence supports its effectiveness in treating olfactory function from various causes and in reducing cognitive impairment.

Despite these findings, there is limited research on whether odor enrichment can serve as a mitigating strategy for dNCR among human populations. To address this gap, we conducted a clinical study to investigate whether odor enrichment could mitigate dNCR in geriatric patients and to explore the relationship between olfactory function and dNCR.

ELIGIBILITY:
Inclusion Criteria:

1. were aged at least 65 years old;
2. were expected a postoperative hospital stay of at least 7 days;
3. had American Society of Anesthesiologist (ASA) class I to II;
4. were native Mandarin speakers;
5. had been referred for a total knee or hip replacement under general anesthesia.

Exclusion Criteria:

1. were prior diagnosed of neurologic diseases by the International Statistical Classification of Diseases and Related Health Problems, 10th Revision (ICD-10);
2. had a history of mental disorders diagnosed using the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
3. had a history of illness or surgery with nasal or sinus;
4. caught cold within one week;
5. impaired vision or auditory function which may affect the assessments;
6. were unwilling to comply with the protocol or procedures;
7. did not pass the Mini-mental State Examination (illiterates get less than 18 points, primary school graduates get less than 20 points, secondary school graduates or higher get less than 24 points) .

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of dNCR | 3 days before surgery (baseline) and 7 days after surgery (follow-up)
  Participants underwent neuropsychological test battery, which referred to International Study Group of Postoperative Cognitive Dysfunction (ISPOCD) test battery and modified according to the characteristics of Chinese patients. The neuropsychological test battery consisted of the Hopkins Verbal Learning Test-Revised (HVLT-R), Brief Visuo-spatial Memory Test-Revised (BVMT-R), Trails Making Test (TMT), Digital Span Test (DST), HVLT-R Delayed Recall Test, HVLT-R Recognition Discrimination Index, BVMT-R Delayed Recall Test, BVMT-R Recognition Discrimination Index and Verbal Fluency Test (VFT). According to the International Study of Perioperative neurocognitive disorder definition, dNCR was diagnosed by calculating the "Z-score".

SECONDARY OUTCOMES:
Olfactory identification ability | 3 days before surgery (baseline) and 7 days after surgery (follow-up)
  Five-odor-olfactory detection arrays were applied to test the odor identification ability of the participants three days before and then about 7 days after the surgery. This test consisted of 5 pen-shaped test sticks without labels containing five odorants including vinegar, banana, mint, rose and coal tar odor. After sniffing each stick, participants should identify each odor freely. The interval between odor presentations was about 30 seconds. The scores ranged from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim MS, Yoon JH, Kim HJ, Yong SW, Hong JM. Olfactory dysfunction is related to postoperative delirium in Parkinson's disease. J Neural Transm (Vienna). 2016 Jun;123(6):589-94. doi: 10.1007/s00702-016-1555-0. Epub 2016 Apr 20. PMID 27098668
- [Background] Brown CH 4th, Morrissey C, Ono M, Yenokyan G, Selnes OA, Walston J, Max L, LaFlam A, Neufeld K, Gottesman RF, Hogue CW. Impaired olfaction and risk of delirium or cognitive decline after cardiac surgery. J Am Geriatr Soc. 2015 Jan;63(1):16-23. doi: 10.1111/jgs.13198. PMID 25597555
- [Background] Zhang C, Han Y, Liu X, Tan H, Dong Y, Zhang Y, Liang F, Zheng H, Crosby G, Culley DJ, Marcantonio ER, Shen Y, Cao JL, Xie Z. Odor Enrichment Attenuates the Anesthesia/Surgery-induced Cognitive Impairment. Ann Surg. 2023 Jun 1;277(6):e1387-e1396. doi: 10.1097/SLA.0000000000005599. Epub 2022 Jul 18. PMID 35848747
- [Background] Pieniak M, Oleszkiewicz A, Avaro V, Calegari F, Hummel T. Olfactory training - Thirteen years of research reviewed. Neurosci Biobehav Rev. 2022 Oct;141:104853. doi: 10.1016/j.neubiorev.2022.104853. Epub 2022 Sep 5. PMID 36064146